CLINICAL TRIAL: NCT02916940
Title: Randomized Controlled Prospective Study on the Injection of Corticoids for the Treatment of Acute Sprains of the Proximal Interphalangeal Joints of the Fingers (Thumb Excluded).
Brief Title: Injection of Corticoids for the Treatment of Acute Sprains of the Proximal Interphalangeal Joints of the Fingers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Socorro ORTIZ, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-Diprophos-IPP
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Sprain
Keywords: sprains of the proximal interphalangeal joints of the long fingers; Diprophos
MeSH Terms: conditions — Sprains and Strains | interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diprophos (Experimental): Patients having had a sprain of the long fingers, within 2 weeks of consultation. This group will receive a single injection of corticoids.
  Interventions: Drug: Diprophos
- Control group (No Intervention): Patients having had a sprain of the long fingers (Eaton classification type I and II), within 2 weeks of consultation. This group will receive the standard of care treatment, without injection of corticoids.

INTERVENTIONS:
Drug: Diprophos — Single subcutaneous injection of Diprophos, in the acute phase.
  Arms: Diprophos

SUMMARY:
There is currently no real consensus on the optimal management of acute sprains of the proximal interphalangeal joint of the long fingers.

The aim of this study is to assess the beneficial effect of an injection of corticosteroids for the treatment of this type of sprain (one single sub-cutaneous injection, in the acute phase). This treatment, if effective, might become the treatment of choice for these types of injuries, instead of a prolonged immobilization or a careful early mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Type I and II and III of the Eaton classification (except if fracture/luxation with more than 50% of the articular surface injured)
* Trauma of one articulation only
* Consultation within 2 weeks of trauma

Exclusion Criteria:

* Patients under 18 years old and over 80 years old
* Pregnant/nursing women
* Eaton classification Type II with a fracture affecting more than 50% of the articular surface, or persistant instability after reduction.
* Open wounds, nerve lesion with sensitive issue and any wound needing a surgical intervention
* Underlying pathologies: rhumatological, neurological, congenital (giving hyperextensive articulations as a result)
* Corticoids allergy
* Infection within the treated zone
* Trauma antecedents at the level of the tendons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Flexion/extension deficit | Baseline (day of kenacort injection)
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer.
Flexion/extension deficit | 7 days after injection
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer.
Flexion/extension deficit | 30 days after injection
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer.
Laxity in hyperextension | Baseline (day of kenacort injection)
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer.
Laxity in hyperextension | 7 days after injection
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer.
Laxity in hyperextension | 30 days after injection
  Evaluation of the maximal amplitude of the articulation, as measured by a goniometer
Diameter of the articulation | Baseline (day of kenacort injection)
  Oedema evaluation. Collateral comparison with the same finger of the other hand: result expressed as a ratio
Diameter of the articulation | 7 days after injection
  Oedema evaluation. Collateral comparison with the same finger of the other hand: result expressed as a ratio
Diameter of the articulation | 30 days after injection
  Oedema evaluation. Collateral comparison with the same finger of the other hand: result expressed as a ratio
Prehension force | Baseline (day of kenacort injection)
  Assessed by a dynamometer (Jamar hydraulic gauge). Result expressed as a ratio with the prehension force of the non-injured hand.
Prehension force | 7 days after injection
  Assessed by a dynamometer (Jamar hydraulic gauge). Result expressed as a ratio with the prehension force of the non-injured hand.
Prehension force | 30 days after injection
  Assessed by a dynamometer (Jamar hydraulic gauge). Result expressed as a ratio with the prehension force of the non-injured hand.

SECONDARY OUTCOMES:
EVA scale | 7 days after injection
  Pain assessment at the level of the volar plate
EVA scale | 30 days after injection
  Pain assessment at the level of the volar plate
Mini-DASH | 7 days after injection
  Assessment of the return to daily life activities or sport activities. Questionnaire of the Disabilities of the Arm, Shoulder and Hand.
Mini-DASH | 30 days after injection
  Assessment of the return to daily life activities or sport activities. Questionnaire of the Disabilities of the Arm, Shoulder and Hand.
Mitchigan Hand Questionnaire | 7 days after injection
  Auto-evaluation of the patient regarding the functionality of his/her articulation
Mitchigan Hand Questionnaire | 30 days after injection
  Auto-evaluation of the patient regarding the functionality of his/her articulation

CONTACTS AND LOCATIONS:
Overall Officials: Nader Chahidi, MD, Study Director — Clinique du Parc Léopold
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - Clinique du Parc Leopold, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freiberg A, Pollard BA, Macdonald MR, Duncan MJ. Management of proximal interphalangeal joint injuries. J Trauma. 1999 Mar;46(3):523-8. doi: 10.1097/00005373-199903000-00033. No abstract available. PMID 10088864
- [Background] Chalmer J, Blakeway M, Adams Z, Milan SJ. Conservative interventions for treating hyperextension injuries of the proximal interphalangeal joints of the fingers. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD009030. doi: 10.1002/14651858.CD009030.pub2. PMID 23450596
- [Background] Paschos NK, Abuhemoud K, Gantsos A, Mitsionis GI, Georgoulis AD. Management of proximal interphalangeal joint hyperextension injuries: a randomized controlled trial. J Hand Surg Am. 2014 Mar;39(3):449-54. doi: 10.1016/j.jhsa.2013.11.038. Epub 2014 Feb 4. PMID 24503231
- [Background] Micev AJ, Saucedo JM, Kalainov DM, Wang L, Ma M, Yaffe MA. Surgical Techniques for Correction of Traumatic Hyperextension Instability of the Proximal Interphalangeal Joint: A Biomechanical Study. J Hand Surg Am. 2015 Aug;40(8):1631-7. doi: 10.1016/j.jhsa.2015.05.011. Epub 2015 Jul 3. PMID 26143967